CLINICAL TRIAL: NCT01917773
Title: Effect of Octreotide on the Colonic Motility in Pediatric Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Indiana University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 1305011397
Record Dates: First submitted 2013-08-02; First posted 2013-08-07 (Estimated); Results first posted 2015-12-21 (Estimated); Last update posted 2015-12-21 (Estimated); Status verified 2015-12

CONDITIONS: Colonic Motility Index; Constipation
MeSH Terms: conditions — Constipation | interventions — Octreotide; Bisacodyl

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Octreotide (Experimental): All patient received octreotide. We compared pre (fasting) and post octreotide colonic motility index.
  Interventions: Drug: Octreotide; Drug: Bisacodyl

INTERVENTIONS:
Drug: Octreotide — Average MI for all patients was calculated over 15-minutes, 30-minutes and 45- minutes before and after administration of octreotide
  Other Names: post octreotide
Drug: Bisacodyl

SUMMARY:
The research study is designed to test how a medication called octreotide affects the motility (contraction or squeezing) of the colon (large intestine). Investigators are investigating whether octreotide can increase contraction and movement in the colon.

DETAILED DESCRIPTION:
As mentioned above.

ELIGIBILITY:
Inclusion Criteria:

* Male or female and undergoing colonic manometry for a routinely accepted indication including: evaluation of chronic constipation, unexplained abdominal distension (Should have had previous diagnostic work up), recurrent fecal impaction, post Hirschsprung's disease repair, chronic intestinal pseudo-obstruction, or suspected colonic dysmotility of any other cause.
* Children aged 12 months or older who are undergoing colonic motility under the supervision of Dr. Joseph Croffie at Riley Hospital.
* In the investigator's judgment, parent(s)/guardian(s) is mentally competent to provide informed consent to participate in the study.

Exclusion Criteria:

* • Subjects with known or suspected allergy to octreotide.

  * Subjects with known prolonged corrected QT interval (QTc) Syndrome or highest risk QTc-Prolonging Agents (including mifepristone).
  * Subjects with known history of ventricular arrhythmia.
  * Subjects with history of any organ transplant who are taking cyclosporine at the time of the motility study.
  * Subjects with history of small bowel transplant.
  * Subjects less than 12 months old.
  * Subjects with severe renal impairment
  * Subjects with severe hepatic impairment
  * Subjects taking bromocriptine, insulin, oral hypoglycemic agents, beta blockers, calcium channel blockers, quinidine, terfenadine, pimozide, sildenafil, tadalafil, and any agents to control fluid and electrolyte imbalance

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 13 (Actual)
Dates: Start 2013-08; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Croffie, Study Director — Riley Hospital for Children
Locations (1):
- Motility Laboratory, Division of Pediatric Gastroenterology, Hepatology and Nutrition at the James Whitcomb Riley Hospital for Children,, Indianapolis, Indiana, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All eligible patients referred for colonic manometry to the GI Motility Laboratory at Riley Hospital between Sep 2013 and June 2014.
  24 patients were assessed for eligibility to participate in the study in the hospital. 8 patients were excluded, as they did not meet inclusion criteria. 3 participant refused enrollment.
Groups:
- Octreotide: This was a non-randomized, single center, open label, and prospective study. Thirteen patients were enrolled in the study. All patient received Octreotide as per study protocol.
Period: Overall Study
Arm/Group | Octreotide
Started | 13
Completed | 13
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Octreotide: 1. Fasting motility was recorded for at least 60 minutes.
  2. Octreotide 1mcg/kg, maximum of 50mcg was administered subcutaneously (one hour after application of EMLA topical cream). Motility was then recorded for 45-60 minutes.
  3. Patients were then offered a high-fat, high-energy meal as described elsewhere, and motility was recorded for 60 minutes.
  4. Patients then received 1 to 2 doses of bisacodyl (0.2 mg/kg, maximum of 10 mg) through the motility catheter, and motility was recorded.
Arm/Group | Octreotide
Number analyzed (Participants) | 13
Age, Continuous [Mean (Full Range); unit: years] | 9.3 [4.6 to 16.2]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 12
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Compared Colonic Motility Index From Fasting to Post Octreotide Infusion
Description: Colonic motility was measured using a solid-state catheter. The catheter had 36 sensors spaced 5-cm apart for the first 15 sensors and 1-cm apart for the remaining sensors. Pressures were transmitted to a transducer and recorded on a personal computer system (Medical Measurement Systems USA, Dover, NH).
  Motility index (MI) was calculated using the Medical Measurement Systems computer program. The MI represents the area under the curve of the pressure tracing for a certain period (21). The MI was calculated for each channel. The MIs from all of the channels were then averaged to give each patient 1 average MI for the particular period under study. In this study, MI was calculated for the periods of 15, 30, and 45 minutes before and after infusion of octreotide. MI is reported as millimeters of mercury (mmHg) per 15, 30, or 45 minutes.
Time Frame: Average MI for all patients was calculated over 15-minutes, 30-minutes and 45- minutes before and after administration of octreotide.
Measure: Mean (95% Confidence Interval); unit: mm Hg
Groups:
- 15 Minutes: The MI for the 15 minutes before and after octreotide infusion was measured.
- 30 Minutes: The MI for the 30 minutes before and after octreotide infusion was measured.
- 45 Minutes: The MI for the 45 minutes before and after octreotide infusion was measured.
Arm/Group | 15 Minutes | 30 Minutes | 45 Minutes
Number analyzed (Participants) | 13 | 13 | 13
mm Hg
  pre-octreotide | 6.03 [5.35 to 6.72] | 6.89 [6.14 to 7.64] | 7.73 [7.01 to 8.45]
  post-octreotide | 5.32 [4.42 to 6.23] | 6.71 [5.91 to 7.52] | 7.53 [6.78 to 8.28]
Statistical Analysis 1: Comparison: 15 Minutes; The Wilcoxon signed rank test was used to analyze change in MI at 15 minutes. Values were considered to be significant if P <0.05; Test type: Non-Inferiority or Equivalence — Reported MIs and SDs in healthy volunteers from an adult study were used to calculate sample size (1). A sample size of 13 patients was deemed adequate to detect a 25% change in MI with 80% power. Reference: Rao SS, Kavelock R, Beaty J, Ackerson K, et al. Effects of fat and carbohydrate meals on colonic motor response. Gut. Feb 2000;46(2):205-211; p = 0.087, Wilcoxon signed rank test
Statistical Analysis 2: Comparison: 30 Minutes; The Wilcoxon signed rank test was used to analyze change in MI at 30 minutes. Values were considered to be significant if P <0.05; Test type: Superiority or Other; p = 0.552, Wilcoxon signed rank test
Statistical Analysis 3: Comparison: 45 Minutes; The Wilcoxon signed rank test was used to analyze change in MI at 45 minutes. Values were considered to be significant if P <0.05; Test type: Superiority or Other; p = 0.807, Wilcoxon signed rank test

ADVERSE EVENTS:
Groups:
- All Patients: All 13 patient received octreotide injection. Motility Index (MI) (mm Hg) for the 15 minutes before and after octreotide infusion was measured.
Arm/Group | All Patients
Serious Adverse Events (participants affected / at risk) | 0/13
Other Adverse Events (participants affected / at risk) | 7/13
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | All Patients (N=13)
Mild discomfort with administration of subcutaneous octreotide (Skin and subcutaneous tissue disorders) | 6
mild abdominal discomfort (Gastrointestinal disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No